CLINICAL TRIAL: NCT04968457
Title: Multicenter Post-marketing Survey of SEBBIN Group Silicone Gel-filled Breast Implants
Acronym: IM02
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe SEBBIN (Industry)
Responsible Party: Sponsor
Other Study IDs: PEC 15-10-001
Record Dates: First submitted 2021-07-06; First posted 2021-07-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Implant; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to allow Groupe SEBBIN to communicate to competent authorities and to the scientific community data relative to the safety and effectiveness of SEBBIN silicone gel-filled breast implants.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18-year-old.
* The patient is genetically a woman.
* The patient is candidate to a breast augmentation or breast reconstruction with silicone gel-filled breast implants.
* The patient gets all information regarding the study and signs the informed consent relative to the use of her personal data.

Exclusion Criteria:

* The patient is pregnant or breastfeeding.
* The patient has silicone implants somewhere else than in the breast.
* The patient was diagnosed with one of the following pathologies:

  * Systemic lupus erythematous, Sjogren syndrome, scleroderma, polymyositis, or any other connective tissue disease.
  * Rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, or any other inflammatory arthritic disease.
  * Arthritis, fibromyalgia, chronic fatigue syndrome, or any other mechanic or degenerative non-inflammatory rheumatic disease.
* The patient has a pathology that could delay healing (does not apply to the reconstruction group).
* The patient has cancer (does not apply to the reconstruction group).
* The patient has anatomical or physiological conditions that could lead to postoperative complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrollment in the study was proposed to women over 18-year who were scheduled for a breast augmentation or breast reconstruction with SEBBIN silicone gel-filled breast implants.
Sampling Method: Non-Probability Sample
Enrollment: 908 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Complication | At 10 years of follow-up
  complication rate